CLINICAL TRIAL: NCT03750734
Title: Target Validation and Discovery in Idiopathic Bronchiectasis
Status: Completed | Type: Observational
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: P02437
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Bronchiectasis; Idiopathic Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — Bronchoscopy; Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, bronchial biopsy, bronchial brushings, bronchoalveolar lavage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Idiopathic bronchiectasis: Idiopathic bronchiectasis participants
  Interventions: Diagnostic Test: Bronchoscopy; Diagnostic Test: Blood test
- Healthy volunteers: Healthy volunteers
  Interventions: Diagnostic Test: Bronchoscopy; Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Bronchoscopy — Flexible bronchoscopy will be performed under sedation (typically a sedative such as intravenous midazolam and/or fentanyl) with local anaesthetic to the throat and vocal cords. Bronchial epithelial tissue (via bronchial brushing and biopsy forceps) and bronchial lavage samples will be taken for analysis.
Diagnostic Test: Blood test — Peripheral blood will be taken to collect peripheral blood monocytes, which will then allow the production of induced pluripotent stem cell derived bronchial epithelial tissues.

SUMMARY:
Bronchiectasis is a long-term lung condition where the airways become abnormally enlarged, leading to a build-up of mucus and inflammation that makes the lungs more susceptible to recurrent infection. Patients with bronchiectasis have subtle abnormalities in the way their airway cells respond to infection that are, in part, responsible for the development of their condition. At present there are no licensed treatments for bronchiectasis.

This study will aim to characterise in depth some of these abnormalities with a view to future studies that will try to develop treatments that can directly target those abnormalities at a molecular level.

Patients known to have bronchiectasis who have provided written informed consent will be enrolled alongside healthy volunteers and patients with chronic obstructive pulmonary disease and cystic fibrosis, for comparison. Participants will give a blood sample and have a bronchoscopy. This is a thin telescopic tube, passed through the nose or mouth, under sedation, into the airways that will allow a sample of bronchial epithelial cells to be taken.

The main objective of the study is to achieve a greater understanding of some of the key biological processes/pathways and disease marker genes that play a role in the development of bronchiectasis. This is important because, at present, little is known about the underlying disease mechanisms and there are no licensed treatments for bronchiectasis.

The investigator's hope this in-depth characterisation of specific bronchial epithelial cell abnormalities in bronchiectasis will shed light on novel targets for future drug discovery.

ELIGIBILITY:
Inclusion Criteria:

Bronchiectasis participants

1. Confirmed HRCT diagnosis of bronchiectasis in more than 1 lobe
2. Bronchiectasis not attributable to another cause, e.g. cystic fibrosis/ABPA/PCD
3. Absence of significant emphysema, COPD or asthma
4. Have provided written informed consent that they are willing to participate in the study prior to sample collection

COPD participants (disease controls)

1. Confirmed diagnosis of COPD according to GOLD (Global Initiative for Chronic Obstructive Lung Disease) criteria (FEV1/FVC ratio < 0.70)
2. Absence of significant bronchiectasis on HRCT
3. Have provided written informed consent that they are willing to participate in the study prior to sample collection

Cystic fibrosis participants (disease controls)

1. Have a confirmed diagnosis of cystic fibrosis
2. Have provided written informed consent that they are willing to participate in the study prior to sample collection

Healthy controls

1. No history or diagnosis of clinically significant lung disease
2. Be a non-smoker for > 1 year at screening and have < 5 pack year history of smoking
3. Have provided written informed consent that they are willing to participate in the study prior to sample collection

Exclusion Criteria:

1. Any clinically significant acute illness, including recent exacerbation of lung disease requiring treatment with oral or intravenous antibiotics, in 6 weeks prior to screening
2. Any contraindication to safe bronchoscopy as judged by CI or clinical team (FEV1 < 30% predicted, oxygen saturations < 92% on room air etc.)
3. Any clinically significant bleeding disorder or use of anticoagulant/antiplatelet therapy that could place participants at risk of bleeding
4. Any contraindication to sedation or local anaesthetic medications used for bronchoscopy
5. Current smoking within 6 months prior to screening (defined as someone who has smoked at least one cigarette per day (or pipe, cigar, or cannabis) for ≥ 30 days within 6 months prior to screening)
6. Acute MI, acute stroke or major surgery within 6 months prior to screening
7. History of uncontrolled ischaemic heart disease that place participants at risk during bronchoscopy
8. History of ventilatory failure or hypercapnia that may complicate bronchoscopy
9. Any known active tuberculous or non-tuberculous mycobacterial infection
10. Any use of oral corticosteroids within 4 weeks of screening
11. Any systemic immunomodulatory or immunosuppressive therapy within 3 months of screening
12. Known current malignancy or current evaluation for a potential malignancy
13. Any other clinically significant medical disease that is uncontrolled despite treatment, that is likely, in the opinion of the investigators, to impact the patient's ability to safely participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Secondary care respiratory clinics
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
Identification and comparison of molecular pathways, including through gene expression analysis of airway tissues. | 2 years
  Identification and comparison of molecular pathways, including through gene expression analysis of airway tissues.

SECONDARY OUTCOMES:
Generation of air liquid interface cultures from primary bronchial epithelial cells/IPSC derived bronchial epithelial cells | 2 years
  Generation of air liquid interface cultures from primary bronchial epithelial cells/IPSC derived bronchial epithelial cells
Functional characterisation of airway epithelium | 2 years
  Functional characterisation of airway epithelium

CONTACTS AND LOCATIONS:
Overall Officials: Dr W Flowers, Principal Investigator — Royal Papworth Hospital
Locations (1):
- Royal Papworth Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No